CLINICAL TRIAL: NCT05802277
Title: Characterization of the Mechanical Properties of the Hamstring Muscle Group in Female Athletes: Impact of the Menstrual Cycle and Adaptations to Exercise.
Brief Title: Characterization of the Mechanical Properties of the Hamstring Muscle Group in Female.
Acronym: MECA_CYCLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EZUS-LYON 1 (Other)
Collaborators: Laboratoire Interuniversitaire de Biologie de la Motricité (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 004B2022
Record Dates: First submitted 2023-03-03; First posted 2023-04-06 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Menstrual Cycle; Oral Contraceptive Use
Keywords: Menstrual cycle; Oral contraception; Muscle mechanical properties; shear wave elastography; Hamstrings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menstrual cycle group (Experimental): Women who are not currently taking any form of hormonal contraception and who present a regular menstrual cycle.
  Interventions: Diagnostic Test: Hamstring muscles function assessment
- Oral contraceptive group (Active Comparator): Women taking a second-generation oral contraceptive estrogen-progestogen pill.
  Interventions: Diagnostic Test: Hamstring muscles function assessment

INTERVENTIONS:
Diagnostic Test: Hamstring muscles function assessment — Ultrasound echographic evaluation of the hamstring muscles during stretching and voluntary contractions, before and after a strenuous physical activity.

SUMMARY:
The goal of this clinical trial is to precise the impact of menstrual cycle and physical activity on the hamstrings muscle function in healthy active women. The main question it aims to answer is : is there a moment of the menstrual cycle when the muscle is better able to recover from a strenuous exercise ? Three appointments will be conducted to evaluate the hamstring muscles at difference moments of the menstrual cycle. Echographic and maximal force production measures will be done.

Researchers will compare these results with a group taking oral contraceptives.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged between 18 and 35 years.
* Subjects who practice at least 2 hours of sport per week with a competitive aim.
* Subject who has not presented any musculo-tendinous pathology to the hamstrings in the last 6 months.
* Subject with no musculoarticular pathology having a prolonged (more than 2 weeks) interruption of sports activities in the last 2 years.
* Subject with no muscular pain or pathology currently.
* Subject with no known cardiac disorders or family history that could present a risk known family history that could present a risk in case of intense physical effort.

physical exertion.

* Subjects not taking any medication, which in the opinion of the that, in the opinion of the coordinating investigator, may interfere with the evaluation of the study criteria.
* Subject able and willing to comply with the protocol and agreeing to give written informed consent.
* Subject affiliated or benefiting from a Social Security plan.

Menstrual cycle group:

* Subject whose last 3 menstrual cycles are of a regular duration (± 4 days maximum difference between 2 consecutive menstrual cycles).
* Subject whose last 3 menstrual cycles are of a duration between 24 and 32 days (including milestones).
* Absence of any contraceptive method likely to modulate the hormonal variations linked to the menstrual cycle.

hormonal variations related to the menstrual cycle, during the duration of the duration of the protocol and during the last 6 months after the participant's inclusion.

the participant. Mechanical contraception such as the diaphragm is permitted.

Oral contraceptive group:

- Taking oral contraception, 2nd generation monophasic pill estrogen-progestin pill (Optilova®, Optidril®, Leeloo®, Minidril®, Ludeal®, Zikiale®, Lovavulo®, Lovapharm®) for at least 6 months.

Exclusion Criteria:

* Subjects with a medical contraindication to intense physical activity.
* Subject with a positive pregnancy test result.
* Subject with a medical or surgical history deemed by the coordinating investigator as being incompatible with the study.
* Subjects under guardianship.
* Subjects in a period of exclusion from another study.
* Decision of the volunteer, whatever the reason.
* Adverse event or effect affecting the safety of the volunteer in the opinion of the coordinating investigator.
* Major deviation from the protocol.
* Illness or injury interfering with the normal course of the protocol.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Hamstring muscles shear wave speed | Length of a menstrual cycle (around on 28 day average)
  Differences according to menstrual cycle phase in hamstring muscles shear wave speed, as measured by ultrasound elastography

SECONDARY OUTCOMES:
Maximal voluntary force production | Length of a menstrual cycle (around on 28 day average)
  Differences according to menstrual cycle phase in maximal voluntary isometric hamstrings force production, as measured by an isokinetic dynamometer
Hamstring muscles thickness | Length of a menstrual cycle (around on 28 day average)
  Differences according to menstrual cycle phase in hamstring muscles thickness, as measured by ultrasound echography.
Hamstring muscles length of fascicles | Length of a menstrual cycle (around on 28 day average)
  Differences according to menstrual cycle phase in hamstring muscles fascicles' length, as measured by ultrasound echography.
Hamstring muscles pennation angle | Length of a menstrual cycle (around on 28 day average)
  Differences according to menstrual cycle phase in hamstring muscles pennation angle, as measured by ultrasound echography.
Hamstring muscles cross sectional area | Length of a menstrual cycle (around on 28 day average)
  Differences according to menstrual cycle phase in hamstring muscles cross sectional area, as measured by ultrasound echography.
Hamstring tendons length | Length of a menstrual cycle (around on 28 day average)
  Differences according to menstrual cycle phase in hamstring tendons length, as measured by ultrasound echography.
Maximal knee joint range of motion | Length of a menstrual cycle (around on 28 day average)
  Measure of the volunteer maximal knee range of motion, the maximum being defined by the volunteer as the greatest hip/leg angle reachable without feeling pain. The process is slowly conducted on an isokinetic ergometer by extending the knee joint (2°/s) until the volunteer reaches her maximal range of motion, at which point the movement is stopped and a security is placed.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Fouré, PhD, Principal Investigator — Université Claude Bernard Lyon 1; Cyril Martin, PhD, Study Director — Université Claude Bernard Lyon 1
Locations (1):
- Laboratoire Interuniversitaire de Biologie de la Motricité, Villeurbanne, Rhône, France

IPD SHARING:
Plan to Share IPD: No